CLINICAL TRIAL: NCT01197105
Title: Clinical Evaluation of a Mouthwash Based on Schinus Terebinthifolius (Aroeira) Used by Children With Gingivitis
Brief Title: Evaluation Study of a Mouthwash Based on Schinus Terebinthifolius to Treat Gingivitis in Children
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Ricardo Dias de Castro, Federal University of Paraiba
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: ACTG 2612
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Gingivitis; Plaque Accumulation
Keywords: gingivitis; schinus terebinthifolius; natural products
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aroeira (Experimental)
  Interventions: Biological: Use of natural product (Schinus terebinthifolius)

INTERVENTIONS:
Biological: Use of natural product (Schinus terebinthifolius) — Mouthwash (0,3125% of schinus terebinthifolius) 10mL per day during 14 days.

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of a mouthwash based on a natural product (Schinus terebinthifolius) used by children with gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 10-12 years old
* Presence of at least 20 dental elements
* Do not use orthodontic fixed appliances
* Simplified Oral Hygiene Index (S-OHI) is greater than 2
* Levels of Microbiological Streptococcus mutans in saliva high (> 10,000 CFU / mL) (JENSEN; BRATTHALL, 1989)
* Susceptibility to form biofilm and gingival inflammation
* Absence of systemic disease
* Not be under the use of antiseptic mouthwash in the last 3 months

Exclusion Criteria:

-

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Gingival inflammation (Blood gingival index) | baseline
  In this time frame will be assessed the initial gingival inflammation in children.
Plaque amount | Baseline
  In this time will be assessed the initial oral hygiene condition of the children before the use of the product through the Simplified Oral Hygiene Index.

SECONDARY OUTCOMES:
Gingival inflammation (Blood gingival Index) | After 7 days (t1)
  In this time frame will be assessed the gingival inflammation in children after 7 days using the product.
Gingival inflammation (blood gingival index) | After 14 days (t2)
  In this time frame will be assessed the final condition of the children after 14 days using the product.
Plaque amount | After 7 days (t1)
  In this time will be assessed the oral hygiene condition of the children after 7 days using the product (Through Simplified Oral Hygiene Index).
Plaque amount | After 14 days (t2)
  In this time will be assessed the final oral hygiene condition of the children after 14 days using the product (through the Simplified Oral Hygiene Index).

CONTACTS AND LOCATIONS:
Locations (1):
- Francisco Campos Statal School, João Pessoa, Paraíba, Brazil

REFERENCES:
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341